CLINICAL TRIAL: NCT03711630
Title: Impact of Meditation on Bothersome Tinnitus
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: State University of New York at Buffalo (Other)
Collaborators: University at Buffalo (Other)
Responsible Party: Principal Investigator, Brendan P. Fitzgerald, Principal Investigator, State University of New York at Buffalo
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: STUDY00002602
Record Dates: First submitted 2018-10-09; First posted 2018-10-18 (Actual); Last update posted 2020-10-22 (Actual); Status verified 2020-10

CONDITIONS: Tinnitus; Noise Induced Tinnitus; Tinnitus, Subjective; Tinnitus, Objective; Tinnitus Aggravated; Tinnitus, Pulsatile; Tinnitus, Spontaneous Oto-Acoustic Emission; Tinnitus, Clicking; Tinnitus, Tensor Tympani Induced
MeSH Terms: conditions — Tinnitus | interventions — Meditation

STUDY DESIGN:
Intervention Model Description: This study is a non-randomized interventional study in which subjects with bothersome tinnitus will meditate to investigate how meditation effects the level of bother of their tinnitus.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Meditation (Experimental): The study cohort will participate in self-guided meditation practice over the course of eight weeks.
  Interventions: Behavioral: Meditation

INTERVENTIONS:
Behavioral: Meditation — Meditation practice will be through the InsightTimer smart device application. Participants will choose what types of meditation practices they will engage in and report their time spent meditating via REDCap.

SUMMARY:
The purpose of this mixed methods correlational study is to investigate the effects of meditation on the level of bother in tinnitus patients in the United States. The researchers seek to understand the changes in bother as compared to the amount of time spent meditating. Data is obtained through the Insight Timer mediation application. Outcome measures will include several validated and reliable measures.

DETAILED DESCRIPTION:
Mindfulness is a practice of "careful attention to mental and physical processes." ("Glossary of Buddhist Terms," 2018) Mindfulness is a component of various types of spiritual practices including meditation, specifically, from Buddhist tradition. While there are many types of meditative activities, Western medicine has begun to focus on practices most closely related to Vipassana Meditation, also known as, Insight Meditation. Mindfulness can be considered a component of meditation practices, but can also be practiced and incorporated in to an individual's daily activity.

While meditation has long been a practice in several Eastern religions and spiritual practices, it most notably came to Europe and North America in the early 1960s. By 1976, the Insight Meditation Society, one of the first retreat centers in the United States, was founded by Joseph Goldstein, Sharon Salzburg, and Jack Kornfield ("Celebrating 40 Years (1976-2016)," 2018). From this, developed the medical research around mindfulness of Jon Kabat-Zinn, Founder of the UMass Medical School Mindfulness Based Stress Reduction (MBSR) Program ("History of MBSR," 2017).

Mindfulness practice has gained popularity as a first line medical intervention for three main reasons. Mindfulness practice is non-invasive, non-pharmacologic, and has no significant side effects (Cebolla, Demarzo, Martins, Soler, & Garcia-Campayo, 2017). Since it is non-invasive, mindfulness on its own is rarely harmful, however, if used in the place of proven interventions can be dangerous. Those utilizing mindfulness practices and meditation must still be under the care of appropriate medical professionals. As a non-pharmacologic intervention, it can be cost effective and not financially prohibitive or burdensome for patients. While the quality of instruction and subsequent practice should be further investigated, the practice itself has the potential to be available at little cost. Much like exercise, meditation and mindfulness practice can be subject to failure if a patient is not compliant to the regimen. Since there is still much to know about the impacts of the types and qualities of meditation on an individual level, its potential benefits can greatly outweigh any risks.

For the purposes of this study meditation and meditative activities will not be limited only to mindfulness, which can be one aspect of meditation. Meditation can be categorized into three areas. Focused attention (FA) or concentration meditation is a practice in which the practitioner focuses their attention on a singular idea or object (Rinpoche, 1980) as in breath awareness, metta or loving-kindness meditation, or a repeated word or phrase as in transcendental meditation. This has typically become a starting point for most novice practitioners. Open-monitoring (OM) includes mindfulness practice, in which the practitioner seeks to become aware of physical and emotional states, responses, and activities. The third category of meditation is one that combines both Focused Attention and Open-monitoring Meditation. This includes Vipassana practice, or Insight meditation, from which Kabat-Zinn has developed the MBSR model. The first two practices rarely are exclusive of each other, but rather, a practitioner's session may include FA and OM.

Previous study of meditation has demonstrated activations and changes in specific regions of the brain. Findings from Manna et al., indicate that expert meditators control cognitive engagement in conscious processing of sensory-related, thought and emotion contents, by massive self-regulation of fronto-parietal and insular areas in the left hemisphere, in a meditation state-dependent fashion. We also found that anterior cingulate and dorsolateral prefrontal cortices play antagonist roles in the executive control of the attention setting in meditation tasks. … Finally, our study suggests that a functional reorganization of brain activity patterns for focused attention and cognitive monitoring takes place with mental practice, and that meditation-related neuroplasticity is crucially associated to a functional reorganization of activity patterns in prefrontal cortex and in the insula. (2010) Others have confirmed through the use of fMRI that meditative methods of MBSR, Mindfulness Cognitive Behavioral Therapy (MCBT), and dispositional mindfulness - the present moment awareness in daily life - change functional and structural components of the prefrontal cortex, cingulate cortex, insula, hippocampus, and amygdala after an eight-week program. These findings indicate emotional and behavioral changes being related to those functional and structural changes (Gotink, Meijboom, Vernooij, Smits, & Hunink, 2016). These changes were found to be similar to those noted in experienced meditators.

Others found changes in functional connectivity in the medial prefrontal cortex, right thalamus/parahippocampal gyrus, and bilateral anterior insula/putamen during meditation. These findings were associated with top-down cognitive, emotion, and attention control in the practice of mental silence in Sahaja Yoga meditation (Hernandez, Barros-Loscertales, Xiao, Gonzalez-Mora, & Rubia, 2018).

A meta-analysis by Merkes of fifteen studies on the effects of MBSR has demonstrated improved functional outcomes for chronic conditions including "fibromyalgia, chronic pain, rheumatoid arthritis, type 2 diabetes, chronic fatigue syndrome, multiple chemical sensitivity, and cardiovascular diagnoses." This analysis also reported no negative outcomes between baseline and follow-up assessments (Merkes, 2010).

While it can be difficult to differentiate and locate the source of a patient's tinnitus, it is thought to originate in any combination of three areas - namely peripherally from the auditory system, centrally, or from somatosensory input. Tinnitus is commonly associated with specific regions of the brain, particularly, the Dorsal Cochlear Nucleus, Central Auditory Pathway, and Auditory Cortex (Han, Lee, Kim, Lim, & Shin, 2009). Most recently, using residual inhibition, Sedley et al. found tinnitus activity in the thalamus, and contrary to expectations, almost all of the auditory cortex and large portions of the temporal, parietal, sensorimotor, and limbic cortex (2015).

Given tinnitus is believed to cause neuroplastic changes in several areas of the brain (Han et al., 2009) and that meditation and mindfulness activities are shown to make restorative changes in those same areas while improving emotional responses, this study investigates the association between the amount of time spent and type of meditation and relief from tinnitus through reduction of bother.

McKenna et al., have found significant reduction of bother in patients with chronic tinnitus through the use of Mindfulness-Based Cognitive Therapy (MBCT), a standardized approach to tinnitus management following an eight-week MBCT program led by clinical psychologists. They rightly point out that much of the current research in non-standardized approaches, like the one proposed in this study, has been limited by small sample sizes (2018). This study looks to add to the body of research for non-standardized interventions and lead to the possibility of increased access to care for patients.

ELIGIBILITY:
Inclusion Criteria:

* Adults, age 18 and above, self-reporting bothersome tinnitus lasting longer than three months.
* Have been evaluated by an audiologist or otologist.

  * Those willing and able to utilize their own smart device or computer meeting the following requirements. For Mac: Requires iOS 10.0 or later. Compatible with iPhone, iPad, and iPod touch.
  * For Android: varies by device.
  * Data and/or Wi-Fi access

Exclusion Criteria:

* Individuals with meditation training or consistent meditation practice (practice that totals more than 20 minutes daily) within the past six months.
* Those indicated by the Hospital Anxiety and Depression Scale to have "abnormal" indications for anxiety or depression.
* Those with any conditions that would restrict them from being able to either sit, walk, or lie down for at least 30 minutes at a time.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 27 (Actual)
Dates: Start 2018-10-06 (Actual); Primary Completion 2019-02-23 (Actual); Study Completion 2020-03-21 (Actual)

PRIMARY OUTCOMES:
Tinnitus Handicap Questionnaire (Change in Bother from Tinnitus Over Time) | Week 1, Week 3, Week 8
  A measure of degree of bother imposed by tinnitus on the patient.

SECONDARY OUTCOMES:
Tinnitus Handicap Inventory | Week 1, Week 3, Week 8
  A measure of degree of bother imposed by tinnitus on the patient.
Hospital Anxiety and Depression Scale | Week 1, Week 3, Week 8
  A scale to determine the degree and impact of a participant's anxiety and depression.
  Scoring:
  Total score: Depression (D) ___________ Anxiety (A) ______________ 0-7 = Normal 8-10 = Borderline abnormal (borderline case) 11-21 = Abnormal (case) 16-21 = exclusionary for participation in this study
Tinnitus Functional Index | Week 1, Week 3, Week 8
  A measure of degree of bother imposed by tinnitus on the patient.
Mindful Attention Awareness Scale | Week 1, Week 3, Week 8
  A measure to determine the degree of mindful attention the participant utilizes in their lives during the course of the study.
  To score the scale, simply compute a mean of the 15 items. Higher scores reflect higher levels of dispositional mindfulness.

CONTACTS AND LOCATIONS:
Locations (1):
- University at Buffalo, Buffalo, New York, United States

IPD SHARING:
Plan to Share IPD: No
This study will not share IPD beyond authors within this study.

REFERENCES:
- [Background] National Health and Nutrition Examination Survey. (2013). Retrieved from https://wwwn.cdc.gov/nchs/nhanes/2011-2012/AUQ_G.htm.
- [Background] Alsubaie M, Abbott R, Dunn B, Dickens C, Keil TF, Henley W, Kuyken W. Mechanisms of action in mindfulness-based cognitive therapy (MBCT) and mindfulness-based stress reduction (MBSR) in people with physical and/or psychological conditions: A systematic review. Clin Psychol Rev. 2017 Jul;55:74-91. doi: 10.1016/j.cpr.2017.04.008. Epub 2017 Apr 23. PMID 28501707
- [Background] Anheyer D, Haller H, Barth J, Lauche R, Dobos G, Cramer H. Mindfulness-Based Stress Reduction for Treating Low Back Pain: A Systematic Review and Meta-analysis. Ann Intern Med. 2017 Jun 6;166(11):799-807. doi: 10.7326/M16-1997. Epub 2017 Apr 25. PMID 28437793
- [Background] Bhatt JM, Lin HW, Bhattacharyya N. Prevalence, Severity, Exposures, and Treatment Patterns of Tinnitus in the United States. JAMA Otolaryngol Head Neck Surg. 2016 Oct 1;142(10):959-965. doi: 10.1001/jamaoto.2016.1700. PMID 27441392
- [Background] Candia V, Wienbruch C, Elbert T, Rockstroh B, Ray W. Effective behavioral treatment of focal hand dystonia in musicians alters somatosensory cortical organization. Proc Natl Acad Sci U S A. 2003 Jun 24;100(13):7942-6. doi: 10.1073/pnas.1231193100. Epub 2003 May 27. PMID 12771383
- [Background] Cebolla A, Demarzo M, Martins P, Soler J, Garcia-Campayo J. Unwanted effects: Is there a negative side of meditation? A multicentre survey. PLoS One. 2017 Sep 5;12(9):e0183137. doi: 10.1371/journal.pone.0183137. eCollection 2017. PMID 28873417
- [Background] Chou R, Deyo R, Friedly J, Skelly A, Hashimoto R, Weimer M, Fu R, Dana T, Kraegel P, Griffin J, Grusing S, Brodt ED. Nonpharmacologic Therapies for Low Back Pain: A Systematic Review for an American College of Physicians Clinical Practice Guideline. Ann Intern Med. 2017 Apr 4;166(7):493-505. doi: 10.7326/M16-2459. Epub 2017 Feb 14. PMID 28192793
- [Background] Gans, J. J., O'Sullivan, P., & Bircheff, V. (2014). Mindfulness Based Tinnitus Stress Reduction Pilot Study A Symptom Perception-Shift Program. Mindfulness, 5(3), 322-333. doi:10.1007/s12671-012-0184-4
- [Background] Goldin P, Ramel W, Gross J. Mindfulness Meditation Training and Self-Referential Processing in Social Anxiety Disorder: Behavioral and Neural Effects. J Cogn Psychother. 2009 Aug;23(3):242-257. doi: 10.1891/0889-8391.23.3.242. PMID 25568592
- [Background] Gotink RA, Meijboom R, Vernooij MW, Smits M, Hunink MG. 8-week Mindfulness Based Stress Reduction induces brain changes similar to traditional long-term meditation practice - A systematic review. Brain Cogn. 2016 Oct;108:32-41. doi: 10.1016/j.bandc.2016.07.001. Epub 2016 Jul 16. PMID 27429096
- [Background] Gotink RA, Younge JO, Wery MF, Utens EMWJ, Michels M, Rizopoulos D, van Rossum LFC, Roos-Hesselink JW, Hunink MMG. Online mindfulness as a promising method to improve exercise capacity in heart disease: 12-month follow-up of a randomized controlled trial. PLoS One. 2017 May 9;12(5):e0175923. doi: 10.1371/journal.pone.0175923. eCollection 2017. PMID 28486559
- [Background] Han BI, Lee HW, Kim TY, Lim JS, Shin KS. Tinnitus: characteristics, causes, mechanisms, and treatments. J Clin Neurol. 2009 Mar;5(1):11-9. doi: 10.3988/jcn.2009.5.1.11. Epub 2009 Mar 31. PMID 19513328
- [Background] Henry JA, Zaugg TL, Myers PJ, Schechter MA. The role of audiologic evaluation in progressive audiologic tinnitus management. Trends Amplif. 2008 Sep;12(3):170-87. doi: 10.1177/1084713808319941. Epub 2008 Jul 15. PMID 18628281
- [Background] Henry JA, Zaugg TL, Schechter MA. Clinical guide for audiologic tinnitus management I: Assessment. Am J Audiol. 2005 Jun;14(1):21-48. doi: 10.1044/1059-0889(2005/004). PMID 16180968
- [Background] Hernandez SE, Barros-Loscertales A, Xiao Y, Gonzalez-Mora JL, Rubia K. Gray Matter and Functional Connectivity in Anterior Cingulate Cortex are Associated with the State of Mental Silence During Sahaja Yoga Meditation. Neuroscience. 2018 Feb 10;371:395-406. doi: 10.1016/j.neuroscience.2017.12.017. Epub 2017 Dec 22. PMID 29275207
- [Background] Jansen EJ, Helleman HW, Dreschler WA, de Laat JA. Noise induced hearing loss and other hearing complaints among musicians of symphony orchestras. Int Arch Occup Environ Health. 2009 Jan;82(2):153-64. doi: 10.1007/s00420-008-0317-1. Epub 2008 Apr 11. PMID 18404276
- [Background] Jayewardene WP, Lohrmann DK, Erbe RG, Torabi MR. Effects of preventive online mindfulness interventions on stress and mindfulness: A meta-analysis of randomized controlled trials. Prev Med Rep. 2016 Nov 14;5:150-159. doi: 10.1016/j.pmedr.2016.11.013. eCollection 2017 Mar. PMID 28050336
- [Background] Lewis JE, Stephens SD, McKenna L. Tinnitus and suicide. Clin Otolaryngol Allied Sci. 1994 Feb;19(1):50-4. doi: 10.1111/j.1365-2273.1994.tb01147.x. PMID 8174302
- [Background] Liu YF, Hu J, Streelman M, Guthrie OW. The epworth sleepiness scale in the assessment of sleep disturbance in veterans with tinnitus. Int J Otolaryngol. 2015;2015:429469. doi: 10.1155/2015/429469. Epub 2015 Jan 8. PMID 25642248
- [Background] Lutz A, Brefczynski-Lewis J, Johnstone T, Davidson RJ. Regulation of the neural circuitry of emotion by compassion meditation: effects of meditative expertise. PLoS One. 2008 Mar 26;3(3):e1897. doi: 10.1371/journal.pone.0001897. PMID 18365029
- [Background] Manna A, Raffone A, Perrucci MG, Nardo D, Ferretti A, Tartaro A, Londei A, Del Gratta C, Belardinelli MO, Romani GL. Neural correlates of focused attention and cognitive monitoring in meditation. Brain Res Bull. 2010 Apr 29;82(1-2):46-56. doi: 10.1016/j.brainresbull.2010.03.001. Epub 2010 Mar 16. PMID 20223285
- [Background] McKenna L, Marks EM, Vogt F. Mindfulness-Based Cognitive Therapy for Chronic Tinnitus: Evaluation of Benefits in a Large Sample of Patients Attending a Tinnitus Clinic. Ear Hear. 2018 Mar/Apr;39(2):359-366. doi: 10.1097/AUD.0000000000000491. PMID 28945659
- [Background] McLean G, Lawrence M, Simpson R, Mercer SW. Mindfulness-based stress reduction in Parkinson's disease: a systematic review. BMC Neurol. 2017 May 15;17(1):92. doi: 10.1186/s12883-017-0876-4. PMID 28506263
- [Background] Merkes M. Mindfulness-based stress reduction for people with chronic diseases. Aust J Prim Health. 2010;16(3):200-10. doi: 10.1071/PY09063. PMID 20815988
- [Background] Newberg AB, Wintering N, Khalsa DS, Roggenkamp H, Waldman MR. Meditation effects on cognitive function and cerebral blood flow in subjects with memory loss: a preliminary study. J Alzheimers Dis. 2010;20(2):517-26. doi: 10.3233/JAD-2010-1391. PMID 20164557
- [Background] Morone NE, Greco CM, Weiner DK. Mindfulness meditation for the treatment of chronic low back pain in older adults: a randomized controlled pilot study. Pain. 2008 Feb;134(3):310-319. doi: 10.1016/j.pain.2007.04.038. Epub 2007 Jun 1. PMID 17544212
- [Background] Park T, Reilly-Spong M, Gross CR. Mindfulness: a systematic review of instruments to measure an emergent patient-reported outcome (PRO). Qual Life Res. 2013 Dec;22(10):2639-59. doi: 10.1007/s11136-013-0395-8. Epub 2013 Mar 29. PMID 23539467
- [Background] Roland LT, Lenze EJ, Hardin FM, Kallogjeri D, Nicklaus J, Wineland AM, Fendell G, Peelle JE, Piccirillo JF. Effects of mindfulness based stress reduction therapy on subjective bother and neural connectivity in chronic tinnitus. Otolaryngol Head Neck Surg. 2015 May;152(5):919-26. doi: 10.1177/0194599815571556. Epub 2015 Feb 24. PMID 25715350
- [Background] Sedley W, Gander PE, Kumar S, Oya H, Kovach CK, Nourski KV, Kawasaki H, Howard MA 3rd, Griffiths TD. Intracranial Mapping of a Cortical Tinnitus System using Residual Inhibition. Curr Biol. 2015 May 4;25(9):1208-14. doi: 10.1016/j.cub.2015.02.075. Epub 2015 Apr 23. PMID 25913402
- [Background] Sizoo BB, Kuiper E. Cognitive behavioural therapy and mindfulness based stress reduction may be equally effective in reducing anxiety and depression in adults with autism spectrum disorders. Res Dev Disabil. 2017 May;64:47-55. doi: 10.1016/j.ridd.2017.03.004. Epub 2017 Mar 22. PMID 28342404
- [Background] Zernicke KA, Campbell TS, Blustein PK, Fung TS, Johnson JA, Bacon SL, Carlson LE. Mindfulness-based stress reduction for the treatment of irritable bowel syndrome symptoms: a randomized wait-list controlled trial. Int J Behav Med. 2013 Sep;20(3):385-96. doi: 10.1007/s12529-012-9241-6. PMID 22618308

DOCUMENTS (1):
  • Study Protocol (2018-09-07): https://cdn.clinicaltrials.gov/large-docs/30/NCT03711630/Prot_000.pdf